CLINICAL TRIAL: NCT06103253
Title: Effect of Intervention With Probiotic on the Gut Microbiota of Healthy Volunteers: a Placebo-controlled Randomized Trial
Brief Title: Effect of Probiotic on the Gut Microbiota of Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023005
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Healthy Adults
Keywords: Probiotics; Gut microbiota; Uric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): a placebo 27 group (maltodextrin)
  Interventions: Dietary Supplement: a Bla80 group
- Probiotic group (Active Comparator): a Bla80 group (maltodextrin + strain BLa80 in 10B /day)
  Interventions: Dietary Supplement: a Bla80 group

INTERVENTIONS:
Dietary Supplement: a Bla80 group — the BLa80 group received 2.9 g of maltodextrin + 0.1 g of BLa80 bacterial powder 10B daily.

SUMMARY:
The goal of this placebo-controlled randomized trial is to test the effect of intervention with Bifidobacterium animalis subsp. lactis BLa80 on the composition of the gut microbiota of healthy volunteers. The main question it aims to answer is whether probiotic can effectively regulate intestinal flora. Participants will take a package of probiotics every day, and their weight was recorded once a week using a weight scale. Blood and stool tests were conducted before and after taking probiotics.

DETAILED DESCRIPTION:
This placebo-controlled study aims to investigate the effect of Bifidobacterium animalis subsp. lactis BLa80 supplementation on the status of the gut microbiota of healthy participants. 112 subjects were randomly divided into a placebo group (maltodextrin) and a Bla80 group (maltodextrin + strain BLa80 in 1 × 10 10 colony-forming units/day). The intervention lasted 8 weeks, and 16S rRNA sequencing technology was used to study the changes in gut microbiota between different groups. Simultaneously, clinical indicators such as alanine transaminase (ALT), aspartate aminotransferase (AST), and uric acid (UC) were measured to illustrate the metabolic effects of BLa80.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 21

Exclusion Criteria:

* Those who have been diagnosed with diabetes or have high blood sugar are not recommended to participate in the test;
* People whose daily diet is too light or too greasy are not recommended to participate in the test; People with special dietary structure caused by weight loss or other reasons (such as ketogenic diet, etc.) are not recommended to participate in the test;
* Other people with special circumstances are not recommended to participate, such as those who are allergic to probiotic products; Pregnant women, breastfeeding women and people under 19 years old and over 45 years old should not be tested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
gut microbiota diversity | 8 weeks
  Before and after taking probiotics, subjects' stool was collected, and stool 16s rRNA was detected by DNA extraction kit.

CONTACTS AND LOCATIONS:
Locations (1):
- National Engineering Laboratory for Deep Processing of wheat and corn, Zhengzhou, Henan, China